CLINICAL TRIAL: NCT02978807
Title: Establishing the Prevalance and Accuracy of Different Diagnostic Techniques for Gestational Diabetes in the Resource-constrained Setting of Eldoret, Kenya
Brief Title: Diagnosis of Gestational Diabetes in Eldoret, Kenya
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Moi University (Other); Purdue University (Other); Indiana Clinical and Translational Sciences Institute (Other)
Responsible Party: Principal Investigator, Sonak Pastakia, Associate Professor, Purdue University
Other Study IDs: 1205008671
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes, Gestational
MeSH Terms: conditions — Diabetes, Gestational | interventions — Point-of-Care Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women between 24 to 32 weeks: Pregnant women with a singleton pregnancy who presented to care between 24 -32 weeks of their pregnancy were included in this study.
  All patients enrolled in the study will receive a random point of care blood sugar, point of care and venous fasting blood sugar, point of care and venous 1 hr/2hr glucose tolerance test, and point of care and venous HbA1c.
  Interventions: Procedure: Point of care and venous screening

INTERVENTIONS:
Procedure: Point of care and venous screening

SUMMARY:
The objective of this study is to determine the most appropriate and effective approach for the diagnosis of gestational diabetes mellitus (GDM) among pregnant women receiving focused antenatal care at Moi Teaching and Referral Hospital (MTRH). This will be done through performing a random blood sugar, fasting blood sugar, 1 hr/2hr glucose tolerance test, and HbA1c on all participants who meet eligibility criteria and provide written, informed consent. The specific research question is: what is the most appropriate screening and diagnostic strategy for patients receiving antenatal care at MTRH?

DETAILED DESCRIPTION:
1.0 Background

Worldwide, 70 million women in the reproductive age have diabetes or impaired glucose tolerance placing them at risk of complications of hyperglycemia in pregnancy. The global prevalence rates of gestational diabetes mellitus (GDM) vary from between 12% and 14% depending on the population studied.(1,2) The estimated prevalence of GDM has been reported in Western (11.6%) and South Africa (3.8% - 8.8%) but because of the lack of published results and consistency in diagnosis, treatment, and outcomes in Eastern Africa, the extent of the problem of GDM is unknown in Kenya.(2) Estimates from these studies in sub-Saharan Africa (SSA) reveal a widely variable prevalence ranging from 2.4% to 14% with different methodologies and populations of different risk categories. This lack of focused investigation on GDM in Kenya is of concern as preliminary,unpublished data from the Kenyan Global Network Study on birth outcomes suggests that 5.5 % of birth weights in Western Kenya are greater than 4000g, suggesting a substantial potential burden of diabetes mellitus (DM) or GDM in this population.(3) Maternal hyperglycemia during pregancy predisposes the offspring to glucose intolerance in the future by fetal programming. (1,4,5) This vicious cycle can influence and perpetuate the incidence and prevalence of diabetes in any population. Infants born to mothers with diabetes experience double the risk of serious injury at birth, triple the likelihood of caeserean delivery and quadruple the incidence of newborn intensive care unit admissions.(6-8) These maternal, fetal, and neonatal morbidities attributable to diabetes in pregnancy can be prevented with early diagnosis of DM and effective treatment. Within the landscape of care in Western Kenya, pregnancy may be the only time a woman presents for medical care. Therefore, pregnancy is an opportune time to have a receptive audience to screen for possible pregestational diabetes, promote health education, and diagnose glucose intolerance as the woman transitions beyond the postnatal period.

MTRH is the second largest referral hospital in Kenya and serves as a referral center for the whole of Western Kenya. Although access to healthcare is limited in rural areas of Kenya, the Antenatal Clinic at the hospital serves up to 12,000 new mothers annually. Screening for GDM in the antenatal clinic at MTRH is currently limited to a routine urinalysis for glucosuria. Sutherland and colleagues found that 11% of an unselected obstetric population of 1418 women had random glucosuria. However, only 1% of those with glucosuria had an abnormal glucose tolerance test.9 Glucosuria is common in pregnancy and has not been shown to correlate with the diagnosis of GDM.

2.0 Rationale and Specific Aims

The use of a routine urinalysis as a screening strategy for GDM is not consistent with any national or international guidelines.(10-13) There is currently no consensus on the best method to screen for GDM in rural settings lacking infrastructure for venous testing. There are a variety of testing strategies which have been predominantly tested in resource-rich settings and are now used as the standard of care worldwide. Unfortunately, these testing strategies have not been validated or implemented in resource-constrained settings like those existing in Western Kenya.(2) In the United Kingdom, there is a general lack of consensus; most centers employ the 75g glucose tolerance test (Sensitivity 29% and Specificity 96% - these values are for the 75g 2hr postprandial random blood sugar and not the glucose tolerance test), others adopt a two-stage protocol, starting with 50g screen, to be followed, if abnormal, with 75-g glucose tolerance test. Also, according to the WHO criteria and ADA guidelines for GDM diagnosis, a random blood sugar >11mmol/L (198 mg/dL) or a fasting blood sugar >7.0mmol/L (126 mg/dL) meets the threshold for diagnosis of GDM.(12) Because of this uncertainty, the International Association of Diabetes and Pregnancy Study Groups (IADPSG) has recently helped provide greater clarity to this issue by issuing suggested guidelines for diagnosing both gestational diabetes and overt diabetes in pregnancy. They recommend the 75gm oral glucose tolerance test and the cutpoints derived from the Hyperglycemia and Adverse Pregnancy Outcomes (HAPO) study for all patients receiving GDM screening.

As suggested in the IADPSG guidelines and an emerging body of literature, there is growing support for the utilization of the glycosylated hemoglobin (HbA1c) in diagnosing diabetes. (16) Lipska and colleagues report that women and people of African-American ethnicity are more likely to be identified with dysglycemia using HgbA1c than by fasting blood glucose. A notable weakness of this study is that it was performed in adults age 70-79 and thus it is unlcear whether HbAIC can be used as a diagnostic tool in pregnancy. None of the currently available studies evaluating the use of A1c's for GDM have included African women.(17-20) Several studies have also raised concerns about the accuracy of HbA1c in African populations as the HbA1c results tend to be higher than those seen in other populations.(21-23) Because of the various approaches that are currently being proposed by the IADPSG guidelines, there is still considerable debate over the appropriate test to employ as they recommend performing a fasting blood sugar, HbA1c, or random plasma glucose on all women during their first prenatal visit. If a diagnosis of diabetes is not made during this assessment, it is recommended that a 75g oral glucose tolerance test is performed during the 24th to 28th week of the pregnancy to test for GDM. By combining the results of several studies they have also analyzed the additive benefits of combining different strategies. Through this investigation they have concluded that analyzing fasting blood sugars alone enabled them to identify 8.3% of the evaluable population, while the 1 hour glucose measurement identified another 5.7%, and 2 hour glucose measurement identified an additional 2.1%. One major limitation of this investigation, however, was that the cohort did not include patients reflective of the rural SSA population the investigators on this trial serve in Western Kenya. This theme is illustrated throughout this background as there is a deficiency of published results regarding GDM in SSA populations.(10) The IADPSG diagnosis approach also assumes that the vast majority of expectant mothers will have frequent contacts with the healthcare system including early prenatal visits and subsequent visits throughout the pregnancy. This trend is not commonly seen in SSA as a large proportion of expectant mothers deliver at home or have only minimal contact with the healthcare system.(2) Because of these dynamics, there is a clear need to simplify the diagnostic approach for GDM while also assessing the relative utility of each of the testing strategies (ie. random blood sugar, fasting blood sugar, 1 hr/2hr glucose tolerance test, and HbA1c).

Through this proposal, the investigators hope to take the first step towards addressing GDM in this setting by assessing the relative effectiveness of point of care testing strategies, in comparison to the gold standard approach of using the 75gm oral glucose tolerance test in a representative understudied population.

ELIGIBILITY:
Inclusion criteria:

* All pregnant women at 24-32 weeks gestation
* Singleton pregnancies

Exclusion Criteria:

* Pre-existing diagnosis of diabetes
* Participants < 18 years of age
* On medications that affect glucose control
* Unable to complete the study protocol
* Unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective cohort study that will be conducted at Moi Teaching and Referral Hospital, Mediheal Hospital, and Uashin Gishu District Hospital Antenatal Clinic in western Kenya
Sampling Method: Non-Probability Sample
Enrollment: 935 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of Gestational Diabetes via venous 75 gm oral glucose tolerance test | Measured between 24-32 weeks of pregnancy
  We determined prevalence of gestational diabetes by utilizing the gold standard testing strategy recommended by IADPSG. This includes the completion of a venous fasting blood sugar, provision of a 75 gm glucose, 1 hr post prandial venous glucose assessment, 2 hour post prandial venous glucose assessment. We recruited 935 patients of which 616 patients returned for the venous testing and completed these tests.

SECONDARY OUTCOMES:
Specificity, Sensitivity, positive predictive value, and negative predictive value of alternative point of care screening strategies | Measured between 24-32 weeks of pregnancy
  On day 1, a capillary blood sample was obtained to perform a point of care (POC) random blood glucose test and glycated hemoglobin. A 50gm glucose load was then administered capillary blood samples were collected after 1-hr All participants were then expected to return the next day (or within 1 week for those unable to follow-up immediately) after having fasted overnight for ≥ 8 hours.
  Day 2 testing procedures included recommended IADPSG testing alongside the analogous POC tests. Capillary and venous blood samples for measurement of POC and plasma fasting glucose, venous HbA1c and a complete blood count with differential was performed. A 75gm glucose load was then administered with capillary and venous blood samples collected at 1-hr and 2-hrs for measurement of POC and plasma glucose levels.
  The sensitivity, specificity, NPV and PPV of each screening strategy was determined using 2 by 2 matrices with the IADPSG criteria for the venous 75gm OGTT as the gold standard reference.

CONTACTS AND LOCATIONS:
Overall Officials: Sonak D Pastakia, PharmD, MPH, Principal Investigator — Purdue University, Moi University, Indiana University

IPD SHARING:
Plan to Share IPD: No
There is no need to send out IPD and only de-identified data was analyzed

REFERENCES:
- [Background] Ryan EA. Diagnosing gestational diabetes. Diabetologia. 2011 Mar;54(3):480-6. doi: 10.1007/s00125-010-2005-4. Epub 2011 Jan 4. PMID 21203743
- [Background] Zeck W, McIntyre HD. Gestational diabetes in rural East Africa: a call to action. J Womens Health (Larchmt). 2008 Apr;17(3):403-11. doi: 10.1089/jwh.2007.0380. PMID 18328010
- [Background] Liechty E. (personal communication). Global Research Network Study Kenya.
- [Background] International Diabetes Federation. Global Guideline on Pregnancy and Diabetes. Brussels: International Diabetes Federation, 2009.
- [Background] Mbanya JC, Motala AA, Sobngwi E, Assah FK, Enoru ST. Diabetes in sub-Saharan Africa. Lancet. 2010 Jun 26;375(9733):2254-66. doi: 10.1016/S0140-6736(10)60550-8. PMID 20609971
- [Background] Berger H, Crane J, Farine D, Armson A, De La Ronde S, Keenan-Lindsay L, Leduc L, Reid G, Van Aerde J; Maternal-Fetal Medicine Committee; Executive and Coundil fo the Society of Obstetricians and Gynaecologists of Canada. RETIRED: Screening for gestational diabetes mellitus. J Obstet Gynaecol Can. 2002 Nov;24(11):894-912. doi: 10.1016/s1701-2163(16)31047-7. English, French. PMID 12417905
- [Background] Boney CM, Verma A, Tucker R, Vohr BR. Metabolic syndrome in childhood: association with birth weight, maternal obesity, and gestational diabetes mellitus. Pediatrics. 2005 Mar;115(3):e290-6. doi: 10.1542/peds.2004-1808. PMID 15741354
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Jovanovic-Peterson L, Bevier W, Peterson CM. The Santa Barbara County Health Care Services program: birth weight change concomitant with screening for and treatment of glucose-intolerance of pregnancy: a potential cost-effective intervention? Am J Perinatol. 1997 Apr;14(4):221-8. doi: 10.1055/s-2007-994131. PMID 9259932
- [Background] Mamabolo RL, Alberts M, Levitt NS, Delemarre-van de Waal HA, Steyn NP. Prevalence of gestational diabetes mellitus and the effect of weight on measures of insulin secretion and insulin resistance in third-trimester pregnant rural women residing in the Central Region of Limpopo Province, South Africa. Diabet Med. 2007 Mar;24(3):233-9. doi: 10.1111/j.1464-5491.2006.02073.x. PMID 17263763
- [Background] Crowther CA, Hiller JE, Moss JR, McPhee AJ, Jeffries WS, Robinson JS; Australian Carbohydrate Intolerance Study in Pregnant Women (ACHOIS) Trial Group. Effect of treatment of gestational diabetes mellitus on pregnancy outcomes. N Engl J Med. 2005 Jun 16;352(24):2477-86. doi: 10.1056/NEJMoa042973. Epub 2005 Jun 12. PMID 15951574
- [Background] Landon MB, Spong CY, Thom E, Carpenter MW, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Lain KY, Sorokin Y, Peaceman AM, Tolosa JE, Anderson GB; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. A multicenter, randomized trial of treatment for mild gestational diabetes. N Engl J Med. 2009 Oct 1;361(14):1339-48. doi: 10.1056/NEJMoa0902430. PMID 19797280
- [Background] Sutherland HW, Stowers JM, McKenzie C. Simplifying the clinical problem of glycosuria in pregnancy. Lancet. 1970 May 23;1(7656):1069-71. doi: 10.1016/s0140-6736(70)92751-0. No abstract available. PMID 4191957
- [Background] International Association of Diabetes and Pregnancy Study Groups Consensus Panel; Metzger BE, Gabbe SG, Persson B, Buchanan TA, Catalano PA, Damm P, Dyer AR, Leiva Ad, Hod M, Kitzmiler JL, Lowe LP, McIntyre HD, Oats JJ, Omori Y, Schmidt MI. International association of diabetes and pregnancy study groups recommendations on the diagnosis and classification of hyperglycemia in pregnancy. Diabetes Care. 2010 Mar;33(3):676-82. doi: 10.2337/dc09-1848. No abstract available. PMID 20190296
- [Background] Ross G. Gestational diabetes. Aust Fam Physician. 2006 Jun;35(6):392-6. PMID 16751853
- [Background] American Diabetes Association. Gestational diabetes mellitus. Diabetes Care. 2004 Jan;27 Suppl 1:S88-90. doi: 10.2337/diacare.27.2007.s88. No abstract available. PMID 14693936
- [Background] Lipska KJ, De Rekeneire N, Van Ness PH, Johnson KC, Kanaya A, Koster A, Strotmeyer ES, Goodpaster BH, Harris T, Gill TM, Inzucchi SE. Identifying dysglycemic states in older adults: implications of the emerging use of hemoglobin A1c. J Clin Endocrinol Metab. 2010 Dec;95(12):5289-95. doi: 10.1210/jc.2010-1171. Epub 2010 Sep 22. PMID 20861123
- [Background] Kirk JK, D'Agostino RB Jr, Bell RA, Passmore LV, Bonds DE, Karter AJ, Narayan KM. Disparities in HbA1c levels between African-American and non-Hispanic white adults with diabetes: a meta-analysis. Diabetes Care. 2006 Sep;29(9):2130-6. doi: 10.2337/dc05-1973. PMID 16936167
- [Background] Holcomb WL Jr, Mostello DJ, Leguizamon GF. African-American women have higher initial HbA1c levels in diabetic pregnancy. Diabetes Care. 2001 Feb;24(2):280-3. doi: 10.2337/diacare.24.2.280. PMID 11213879
- [Background] Katon J, Williams MA, Reiber G, Miller E. Antepartum A1C, maternal diabetes outcomes, and selected offspring outcomes: an epidemiological review. Paediatr Perinat Epidemiol. 2011 May;25(3):265-76. doi: 10.1111/j.1365-3016.2011.01195.x. Epub 2011 Mar 21. PMID 21470266
- [Background] Sapienza AD, Francisco RP, Trindade TC, Zugaib M. Factors predicting the need for insulin therapy in patients with gestational diabetes mellitus. Diabetes Res Clin Pract. 2010 Apr;88(1):81-6. doi: 10.1016/j.diabres.2009.12.023. Epub 2010 Jan 13. PMID 20071050
- [Background] Brown CJ, Dawson A, Dodds R, Gamsu H, Gillmer M, Hall M, Hounsome B, Knopfler A, Ostler J, Peacock I, Rothman D, Steel J. Report of the Pregnancy and Neonatal Care Group. Diabet Med. 1996 Sep;13(9 Suppl 4):S43-53. No abstract available. PMID 8894455
- [Background] Maegawa Y, Sugiyama T, Kusaka H, Mitao M, Toyoda N. Screening tests for gestational diabetes in Japan in the 1st and 2nd trimester of pregnancy. Diabetes Res Clin Pract. 2003 Oct;62(1):47-53. doi: 10.1016/s0168-8227(03)00146-3. PMID 14581157
- [Derived] Pastakia SD, Njuguna B, Onyango BA, Washington S, Christoffersen-Deb A, Kosgei WK, Saravanan P. Prevalence of gestational diabetes mellitus based on various screening strategies in western Kenya: a prospective comparison of point of care diagnostic methods. BMC Pregnancy Childbirth. 2017 Jul 14;17(1):226. doi: 10.1186/s12884-017-1415-4. PMID 28705184